CLINICAL TRIAL: NCT02356133
Title: The Relationship Among rSO2, MAP,CAM Value, Vital Organ Disfunction and the Outcome of Patients After Operation by Near-Infrared Spectroscopy in Endovascular Neurosurgery
Brief Title: The Relationship Among rSO2, MAP, et al by Near-Infrared Spectroscopy in Endovascular Neurosurgery
Status: Completed | Type: Observational
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Other Study IDs: 0810-758
Record Dates: First submitted 2015-01-24; First posted 2015-02-05 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Near-Infrared Spectroscopy in Endovascular Neurosurgery
Keywords: Near-Infrared Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
record,describe and discuss the relationship among rSO2, MAP,CAM value, vital organ disfunction and the outcome of patients after operation by Near-Infrared Spectroscopy in Endovascular Neurosurgery

DETAILED DESCRIPTION:
record,describe and discuss the relationship among rSO2, MAP,CAM value, vital organ disfunction and the outcome of patients after operation using Near-Infrared Spectroscopy in Endovascular Neurosurgery meanwhile detect the Brain oxygen supply and function monitoring using noninvasive Near-Infrared Spectroscopy in Endovascular Neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) class I~Ⅲ, ranging in age from 18 to 80 years

Exclusion Criteria:

* ASA>Ⅳ
* Non-cooperators
* Morbid obesity (BMI>35kg/m2)
* Preoperative hyperresponsiveness airway and gastro-esophageal reflux
* The existence of the state or a diagnosis of dementia, delirium, depression, cognitive dysfunction before surgery were also excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Scheduled to undergoing Endovascular Neurosurgery
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
there is relationship between rSO2 and MAP during neurosurgery | 2 month
there is relatinship between rSO2 and CAM values | 2 month
vital organ disfunction related to rSO2 and bad outcome of the patients | 3 month

REFERENCES:
- [Derived] Wang X, Feng K, Liu H, Liu Y, Ye M, Zhao G, Wang T. Regional cerebral oxygen saturation and postoperative delirium in endovascular surgery: a prospective cohort study. Trials. 2019 Aug 14;20(1):504. doi: 10.1186/s13063-019-3586-y. PMID 31412906